CLINICAL TRIAL: NCT04080934
Title: Breaststroke Swimming After Breast Cancer Treatment/Surgery as a Means of Treatment for Seroma, Lymphedema, and Chronic Arm and Chest Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other); Bruyère Health Research Institute. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190304-01H
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Lymphedema; Seroma; Pain, Postoperative; Pain, Chest
MeSH Terms: conditions — Lymphedema; Seroma; Pain, Postoperative; Chest Pain | interventions — Swimming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In the experimental group, patients allocated to the swimming/experimental group will participate in 8 weeks of the swimming program, which involves three weekly swimming sessions of 30 minutes minimum. They will be asked to undergo a range of motion (ROM) assessment by a registered kinesiologist, as well as a few short questionnaires administered over the phone by a research assistant, once at the onset of the intervention and once a month for 3 months during the intervention.
  Interventions: Behavioral: Swimming
- Control Group (No Intervention): The control group will include patients who receive standard of care. This includes the recommendation to undertake exercise and physiotherapy; however, no formal exercise program will be provided. In the control group, participants will be asked to answer a few short questionnaires administered over the phone by a research assistant once per month for 4 months.

INTERVENTIONS:
Behavioral: Swimming — Patients will participate in 8 weeks of the swimming program, which involves three weekly swimming sessions of 30 minutes minimum.
  Arms: Experimental Group

SUMMARY:
Following surgery and treatment for breast cancer, many patients experience swelling of lymph nodes (lymphedema) or accumulation of fluid (seroma) that can cause pain, restrict movement, and reduce quality of life. Current treatments include massage, pressure dressings, and drainage, but these are often ineffective and do not last. Physical activity, in particular swimming, has been linked to improvement in lymphedema/seroma symptoms, but more research is required to determine whether or not this type of treatment is effective.

DETAILED DESCRIPTION:
In 2016, an estimated 25,700 Canadian women were diagnosed with breast cancer. With advances in detection, management and treatment, the 5-year relative survival has improved to 87%. Consequently, breast cancer survivors represent a significant proportion of Canadian society. Research suggests that 30-60 % of women with breast cancer will experience some form of arm morbidity between 6 months and 3 years after breast cancer. Both lymphedema and seroma can cause substantial discomfort, chronic pain, mobility issues, and psychological distress, such as social isolation, anxiety and depression. The current treatment for seroma and lymphedema is drainage, massage, and the use of compression dressings, but these can be ineffective and costly and the effects of the treatment do not last over time. This project will provide crucial knowledge regarding the utility of a simple, swimming based exercise regimen involving the breaststroke in reducing chronic pain related to post-surgical lymphedema or seroma in breast cancer patients. The breaststroke uses a full range of motion in the water, with the water creating a pressure back onto the seroma/damaged tissues. This study will be a randomized, two-arm, pilot study. Patients allocated to the swimming group will participate in 8 weeks of the swimming program, which involves three weekly swimming sessions of 30 minutes minimum. The control group will include patients who receive standard of care. This includes the recommendation to undertake exercise and physiotherapy; however, no formal exercise program will be provided. Breast cancer survivors represent a significant proportion of Canadian society, with most recent data suggesting that at least 157,000 Canadian women who had a breast cancer diagnosis in 1999 were still living. Many of these women still suffer from long term complications of their cancer and its treatment. Given the high prevalence of chronic pain in breast cancer survivors, it is unsurprising that the use of pain medications is prevalent as well. A recent U.S. analysis of 10,000 breast cancer patients treated with adjuvant endocrine therapy demonstrated a 56.9% crude probability of opioid use. Within the context of the current opioid crisis in North America, the opportunity to reduce pain and the need for pain medication is absolutely critical.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants include adult female patients, 18 years of age or higher, from the Ottawa Hospital who are post-operative from a lumpectomy or a mastectomy with or without full axillary dissection and radiation. They will be less than 3 years from completion of their acute cancer treatment. Study subjects must have pain symptoms related to chest wall pain and/or arm morbidity, seroma or lymphedema. They must have approval from their medical and radiation oncologist to participate in the study upon enrollment.

Exclusion Criteria:

* Patients with ongoing medical problems where swimming would be contraindicated will be excluded from this study. Those who swam on a regular basis prior to their breast cancer diagnosis will be excluded from the study, as well as those who cannot swim, due to safety concerns and limited resources/time required to complete more in-depth swimming instruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-08-21 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain following breast cancer | The primary measure will be calculated after swimming is completed. This will last approximately 14 months.
  The primary outcome will be pain as assessed using a visual analog scale (VAS). The VAS scale is a 100mm-long horizontal line with the word "no pain" at one end and "pain as bad as it can be" at the other. This will be pain levels of patients after the swimming program in comparison with the control group who will receive no swimming program.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Mills, MD, Principal Investigator — Univeristy of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No